CLINICAL TRIAL: NCT01621282
Title: Effect of Education on Running Successful Journal Club
Brief Title: Running Successful Journal Club
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nazila zarghi, principal investigator, Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Education
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-06

CONDITIONS: Educational Course
Keywords: journal club
MeSH Terms: interventions — Educational Status; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Experimental): Departments passed 6-month interactive educational course
  Interventions: Other: Education
- No Education (No Intervention): Departments not passed 6-month interactive educational course
  Interventions: Other: Conventional

INTERVENTIONS:
Other: Education — A 6-month interactive course on critical appraisal
  Arms: Education
Other: Conventional — Conventional method/no intervention
  Arms: No Education

SUMMARY:
Running successful journal club is of the important goals for postgraduate education.In this study, the effect of a 6-month interactive educational course on journal clubs of Mashhad Dental school was observed using a valid and reliable checklist(r=0.74). Data will be evaluated and compared using spss software by t-test.

ELIGIBILITY:
Inclusion Criteria:

* Faculty members of Dental School,Postgraduate departments

Exclusion Criteria:

* Faculty members of other schools,Undergraduate departments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
checklist mean score | up to 6 months
  The outcome mesures will be completed up to 6 months